CLINICAL TRIAL: NCT00924040
Title: Retreatment Protocol for BL22 Immunotherapy in Relapsed or Refractory Hairy Cell Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The supply of BL22 has expired and MedImmune the sponsor is not interested in producing any new supply.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Kreitman, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090076; 09-C-0076; NCT00850525 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Hairy Cell Leukemia
Keywords: BL22 in HCL after Immunotoxin; Hairy Cell Leukemia; Leukemia
MeSH Terms: conditions — Leukemia, Hairy Cell; Leukemia | interventions — RFB4(dsFv)-PE38 recombinant immunotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BL22 Immunotherapy (Experimental): 30 micrograms/kg intravenous over 30 minutes every other day (QOD) on days 1, 3, 5, of a 4 week cycle (at least 26 days) for a maximum of 16 cycles or until they become ineligible.
  Interventions: Drug: BL22 (CAT-3888)

INTERVENTIONS:
Drug: BL22 (CAT-3888) — 30 micrograms/kg intravenous over 30 minutes every other day (QOD) on days 1, 3, 5, of a 4 week cycle (at least 26 days) for a maximum of 16 cycles or until they become ineligible.

SUMMARY:
BL22 is a type of protein that scientists have created to interact with certain cancer cells. Experiments have shown that BL22 can bind with cancer cells that have a particular kind of protein (called CD22 ) on their surface, and can kill those cells. CD22 is present on certain types of hairy cell leukemia (HCL) cancer cells, and researchers have been working on treatments that will use BL22 and other related proteins to interact with and kill these kinds of cancer cells. The primary purpose of this study will be to provide access to and treatment with BL22 for patients who have HCL in order to determine their response to the treatment. In addition, the study will assess potential side effects of BL22 and examine why some patients respond better than others to treatment with BL22 and related therapies.

This study will include about 21 to 25 adults who have been diagnosed with forms of HCL that have not responded well to standard treatments such as surgery, chemotherapy, or radiation therapy. These adults also will have received anti-CD22 therapies before, potentially including treatments with BL22, and have not developed immunity or resistance to these treatments.

Prior to the study, patients will undergo a 1- to 2-week screening period to assess their eligibility for treatment. Eligible patients will participate in the study for up to 16 cycles of treatment, with each cycle lasting approximately 4 weeks. For each cycle, patients will receive 1 prescribed dose of BL22 every other day for a total of 3 doses per cycle, and will be assessed after every cycle to evaluate the success of the treatment. During the evaluation visits, patients will be required to have a brief physical examination, give blood and urine samples for testing, and undergo other tests as need to check heart and kidney function and assess the state of the leukemia. Patients who agree will give additional blood, urine, or bone marrow samples for future research purposes.

DETAILED DESCRIPTION:
Background:

BL22, also called CAT-3888 or RFB4(dsFv)-PE38, is a recombinant immunotoxin containing an Fv fragment of an anti-CD22 monoclonal antibody and truncated Pseudomonas exotoxin (PE).

In Phase 1 and 2 trials in patients with chemoresistant hairy cell leukemia (HCL), BL22 showed 47-61% complete remission (CR) rates and 12% of HCL patients had a completely reversible hemolytic uremic syndrome (HUS).

A mutant of BL22, termed CAT-8015 or HA22, differs by 3 amino acids and has higher binding affinity to CD22 compared to BL22 (15-fold greater). CAT-8015 is currently undergoing Phase 1 testing in HCL and other diseases.

HCL patients who have previously received recombinant anti-CD22 immunotoxin (BL22, CAT-8015, or LMB-2) may benefit from additional BL22 administration.

Objectives:

The primary objective is to provide access to BL22 for HCL patients who have previously received BL22, CAT-8015, or LMB-2, or are ineligible for CAT-8015, but may benefit from BL22. The primary outcome will be response to treatment.

Secondary objectives:

* Determine immunogenicity and safety profiles of BL22 in patients with prior immunotoxin, using aspirin/enoxaparin to prevent HUS.
* To correlate response to ex vivo sensitivity of HCL cells, obtained from blood with or without apheresis, to BL22 and to other recombinant anti-CD22 immunotoxins such as CAT-8015, and to tumor markers.
* To correlate neutralizing antibodies with number of cycles of BL22, type and number of prior systemic therapies, and time since prior purine analog.
* To correlate CR by bone marrow biopsy with improvement in bone marrow as assessed by magnetic resonance imaging (MRI) of the spine.

Eligibility:

Patient must have received prior recombinant anti-CD22 immunotoxin (i.e. BL22, CAT-8015, or LMB-2 treatment) or be ineligible for CAT-8015.

HCL with cytopenia, high malignant count or symptomatic splenomegaly.

Patients must have had at least 2 prior systemic therapies. There must have been at least 2 prior courses of purine analog, or 1 if the response to this course lasted < 2 years, or if the patient had unacceptable toxicity to purine analog.

Design:

This is a single institution, expanded access protocol accruing 21-25 patients.

Patients will be administered BL22 at 30 microg/kg every other day for 3 doses (QOD times 3) per 4-week cycle (at least 26 days) for a maximum of 16 cycles.

Patients in CR may receive up to 2 more cycles if without minimal residual disease (MRD), or 4 more cycles if in CR with MRD, but no more than 16 cycles total.

No retreatment if high levels of neutralizing antibodies or progressive disease.

Patients who have been off treatment and relapse after greater than 2 months of a CR or partial response may be retreated if eligibility criteria are still met.

If any HUS, accrual to the study will be suspended for discussion with FDA.

ELIGIBILITY:
* INCLUSION CRITERIA:

One of the following:

1. Patients who previously received CAT-3888 and did not have unacceptable toxicity
2. Patients who received CAT 8015 in study CAT 8015-1001 and have progression of disease or relapse. These patients must be considered off-study for CAT-8015 protocol specified follow-up

Patient must have histopathological evidence of HCL as confirmed by the Laboratory of Pathology, NCI.

At least one of the following indications for treatment:

1. Neutropenia (absolute neutrophil count (ANC) less than 1000 cells/microL).
2. Anemia (hemoglobin (Hgb) less than 10 g/dL).
3. Thrombocytopenia (platelet (Plt) less than 100,000/microL).
4. Absolute lymphocyte count of greater than 5000 cells/microL
5. Symptomatic splenomegaly.
6. Enlarging lymph nodes greater than 2cm.

Patient must have had at least 2 prior systemic therapies. There must have been at least 2 prior courses of purine analog, or 1 if the response to this course lasted less than 2 years, or if the patient had unacceptable toxicity to purine analog.

Patient must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2, unless due to potentially reversible active uncontrolled infection.

Patient must be greater than or equal to 18 years old.

Patient can understand and give informed consent.

Patient must have adequate liver and renal function, as defined by the following criteria:

1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 2.5-times the upper limits of normal.
2. Albumin greater than or equal to 3.0 g/dL.
3. Total bilirubin less than or equal to 2.2 mg/dL.
4. Creatinine less than or equal to 1.4 mg/dL or creatinine clearance greater than or equal to 50 mL/min.

Patient must agree to using adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of the study.

EXCLUSION CRITERIA:

Patients who are pregnant or nursing. A negative pregnancy test (urine or serum) must be documented within one week prior to starting BL22 in women of child-bearing potential.

Patient has developed antibody titer that neutralizes greater than 75% of the activity of 1 microg/mL of BL22 using a bioassay.

Patients who had systemic cytotoxic chemotherapy, immunotherapy, recombinant anti-CD22 immunotoxin (ie, CAT-8015, BL22, or LMB-2) or systemic steroid (with the exception of stable doses of Prednisone less than or equal to 20 mg/day) treatment within 4 weeks of enrollment. Patients receiving a limited number of doses (less than 5) of steroid for non-treatment reasons (eg, allergy prophylaxis connected with medical testing) may not receive any steroid within one week of enrollment and may not have had any evidence of disease response to steroid. Subjects who are receiving steroids for other conditions (e.g., autoimmune disorders) are eligible, as long as there is no increase in the dose or change in steroid type within 1 week of treatment. Subjects who are using a chronic steroid must wait for 4 weeks before starting the trial.

Patient had monoclonal antibody therapy (with the exception of BL22 or CAT-8015 or LMB-2) within 4 weeks of enrollment.

Patient is receiving any other investigational agent.

Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Patients who discontinued from CAT-8015 or BL22 studies due to toxicity or dose-limiting toxicity.

Dose limiting toxicity to CAT-8015

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kreitman, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] BOURONCLE BA, WISEMAN BK, DOAN CA. Leukemic reticuloendotheliosis. Blood. 1958 Jul;13(7):609-30. No abstract available. PMID 13560561
- [Background] Frassoldati A, Lamparelli T, Federico M, Annino L, Capnist G, Pagnucco G, Dini E, Resegotti L, Damasio EE, Silingardi V. Hairy cell leukemia: a clinical review based on 725 cases of the Italian Cooperative Group (ICGHCL). Italian Cooperative Group for Hairy Cell Leukemia. Leuk Lymphoma. 1994 Apr;13(3-4):307-16. doi: 10.3109/10428199409056295. PMID 7519510
- [Background] Vardiman JW, Golomb HM. Autopsy findings in hairy cell leukemia. Semin Oncol. 1984 Dec;11(4):370-80. PMID 6505704
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: United States Food and Drug Administration Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks
- See also: CTCAE — http://ctep.cancer.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed to enroll 21 patients with an expected accrual of 2-3 patients every 2-3 months. Accrual ceiling was 25 patients.
Period: Overall Study
Arm/Group | BL22 Immunotherapy
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BL22 Immunotherapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Months to Response to Treatment
Description: Response is defined by the Response Evaluation Criteria in the protocol, namely the earliest point where all relevant tests (i.e. lab tests, physical exam, radiology results) are consistent with complete response (CR) or partial response (PR). CR or PR must be confirmed for at least 4 weeks. Complete response: No evidence of leukemic cells by routine H/E stains of the peripheral blood and bone marrow. Partial response:neutrophils >/= 1,500/micrograms/L or 50% improvement over baseline without growth factors for at least 4 weeks.
Time Frame: 2/14/2009 till 6/24/2010
Measure: Number; unit: Months
Arm/Group | BL22 Immunotherapy
Number analyzed (Participants) | 1
Months | 2

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 2 years & 6 months
Measure: Number; unit: Participants
Arm/Group | BL22 Immunotherapy
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Number of Participants With Complete Response (CR) Who Resolve the Bone Marrow Abnormality by Magnetic Resonance Imaging (MRI)
Description: Patients are assessed by MRI to determine which ones resolve their marrow abnormality. A non-parametric Wilcoxon test was to be used to determine whether CR correlated with resolution of MRI abnormality
Time Frame: Bone marrow biopsy and MRI 4 weeks after patients meeting blood criteria for CR, and if CR is present, repeat bone marrow biopsy and MRI every 12 months. Bone marrow biopsy and MRI is not done in patients with PR as best response.
Measure: Number; unit: Participants
Arm/Group | BL22 Immunotherapy
Number analyzed (Participants) | 1
Participants | 0

4. Secondary Outcome: Number of Patients Who Developed Neutralizing Antibodies After One or More Cycles of BL22
Description: Fresh malignant cells are isolated from blood, bone marrow, lymph nodes or other tissue and incubated with recombinant immunotoxins to determine sensitivity to BL22 and other agents to estimate the amount of cancer cells in the body by measuring proteins which fall off cancer cells and go into the blood.
Time Frame: 24 weeks
Measure: Number; unit: Participants
Arm/Group | BL22 Immunotherapy
Number analyzed (Participants) | 1
Participants | 0

5. Secondary Outcome: Number of Patients With ex Vivo Sensitivity Who Respond Clinically
Description: Although some hairy cell leukemia (HCL) cells from some patients may have ex vivo sensitivity, they might not respond clinically. Number of participants with pretreatment ex vivo sensitivity (<10 ng/ml IC50) who go on to achieve CR as best response. CR required abscence of HCL in the bone marrow and resolution of cytopenias.
Time Frame: Time to CR can be between 2 months and 1 year
Measure: Number; unit: Participants
Arm/Group | BL22 Immunotherapy
Number analyzed (Participants) | 1
Participants | 0

6. Secondary Outcome: Percentage of Patients Who Respond Clinically, Who Also Have Normalization in sCD22 or sCD25
Description: CD25 (sCD25)and CD22 (sCD22) quantify hairy cell leukemia (HCL) tumor burden. Patients with either PR or CR are evaluated for soluble forms of CD25 (sCD25) and soluble CD22 (sCD22). The number of patients with PR or CR who have normalization of sCD25 and sCD22 will be recorded. Normalization is considered <3 ng/ml for sCD25, and <2 ng/ml for sCD22. Patients will be assessed for normalization of sCD25 and sCD22 for at least 12 months after achieving PR or CR.
Time Frame: patients may undergo lymphapheresis before the first and/or later cycles up to 12 months after achieving CR or PR
Measure: Number; unit: Percentage of participants
Arm/Group | BL22 Immunotherapy
Number analyzed (Participants) | 1
Percentage of participants | 100

7. Secondary Outcome: Correlation Between Number of Prior Cycles of BL22 With Immunogenicity on This Protocol
Description: Percent of patients neutralizing >75% of 1000 ng/ml of BL22 in a biologic assay by end of treatment, with respect to the number of prior cycles of BL22 prior to entry on this protocol
Time Frame: Within 2 months of end of treatment ( measure antibodies before each cycle)
Measure: Number; unit: correlation coefficient
Arm/Group | BL22 Immunotherapy
Number analyzed (Participants) | 1
correlation coefficient | 0

8. Secondary Outcome: Percentage of Patients Who Make Antibodies
Description: Determination of antibodies against BL22 is determined by the Clinical Laboratory Improvement Amendments (CLIA) certified blood tests in our contract lab. NCI-Frederick in the laboratory of Dr. David Waters (Science Applications International Corporation (SAIC). He is CLIA certified.
Time Frame: 24 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | BL22 Immunotherapy
Number analyzed (Participants) | 1
Percentage of participants | 0

9. Secondary Outcome: Percentage of Patients Who Have Dose Limiting Toxicity (DLT)
Description: Determination of dose limiting toxicity (DLT) is by the standard toxicity assessment Common Terminology Criteria for Adverse Events version 3.0 (CTCAEv3.0) done every cycle. For detailed information about the CTCAEv3.0 see the protocol Link module.
Time Frame: 24 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | BL22 Immunotherapy
Number analyzed (Participants) | 1
Percentage of participants | 0

ADVERSE EVENTS:
Arm/Group | BL22 Immunotherapy
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BL22 Immunotherapy (N=1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (4)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1 (2)
Albumin, serum-low (hypoalbuminemia) (Investigations) | 1 (3)
Constipation (Gastrointestinal disorders) | 1 (2)
Constitutional Symptoms - Other (Specify, __) (Nervous system disorders) | 1 (1) — Lightheadedness
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 1 (1) — Rash, tick bite
Diarrhea (Gastrointestinal disorders) | 1 (2)
Edema: limb (General disorders) | 1 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (2)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (4)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Investigations) | 1 (3)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bladder (urinary) (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Leukocytes (total WBC) (Investigations) | 1 (14)
Lipase (Investigations) | 1 (2)
Lymphopenia (Investigations) | 1 (11)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (4)
Metabolic/Laboratory - Other (Specify, __) (Metabolism and nutrition disorders) | 1 (2) — Hypercholesteremia
Pain::Back (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain::Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Platelets (Investigations) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (2)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study of BL22 has expired and MedImmune, the sponsor, is not interested in producing any new supply. All data has been analyzed and reviewed. All patients have been taken off study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No